CLINICAL TRIAL: NCT01192178
Title: A Randomized, Double-Blind, Parallel Group Study of ADVAIR™ DISKUS™ 100/50 and FLOVENT™DISKUS™ 100, Both Twice Daily, in a Pediatric Population During the Fall Viral Season.
Brief Title: Fall Epidemic Viral Pediatric Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 113872
Record Dates: First submitted 2010-07-15; First posted 2010-08-31 (Estimated); Results first posted 2011-11-03 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
Keywords: pediatric; exacerbation; viral induced exacerbation; asthma
MeSH Terms: conditions — Asthma | interventions — BID protein, human; Fluticasone; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FLOVENT™ DISKUS™ 100 mcg (Active Comparator): FLOVENT™ DISKUS™ 100 mcg is an inhaled corticosteroid indicated in the US for maintenance treatment of asthma as prophylactic therapy in patients 4 years and older.
  Interventions: Drug: FLOVENT™ DISKUS™ 100 mcg BID
- ADVAIR™ DISKUS™ 100/50 mcg (Experimental): ADVAIR™ DISKUS™ 100/50 mcg is a combination product containing a corticosteroid and a long acting beta2 adrenergic agonist indicated for; maintenance treatment of asthma in patients 4 years of age and older.
  Interventions: Drug: ADVAIR™ DISKUS™ 100/50 mcg BID

INTERVENTIONS:
Drug: FLOVENT™ DISKUS™ 100 mcg BID — FLOVENT™ DISKUS™ 100 mcg, one inhalation twice daily (BID) from the DISKUS device from randomization through the end of study (week 16).
  Other Names: Fluticasone propionate
  Arms: FLOVENT™ DISKUS™ 100 mcg
Drug: ADVAIR™ DISKUS™ 100/50 mcg BID — ADVAIR™ DISKUS™ 100/50 mcg is a combination product containing a 100 mcg fluticasone propionate and a 50 mcg salmeterol. One inhalation from the DISKUS device twice daily (BID) from randomization through end of study (week 16).
  Other Names: Fluticasone propionate/salmeterol combination
  Arms: ADVAIR™ DISKUS™ 100/50 mcg

SUMMARY:
Study ADA113872 is an exploratory 16-week multi-centre, randomized, double-blind, parallel group study in pediatric subjects, 4 to 11 years of age, with a history of seasonal asthma exacerbation(s). Approximately 40 clinical sites in the United States will randomize 316 subjects. Eligible subjects will be randomly assigned to one of two double-blind treatments using a 1:1 randomization. Subjects will be identified for their eligibility for enrolment starting in April 2010. Eligible subjects will be invited to return for randomization into the study in August 2010. This exploratory study is being conducted to assess whether treatment with ADVAIR™ DISKUS™ 100/50 mcg is more effective at reducing the risk of exacerbation and the asthma impairment associated with viral respiratory tract infections during the fall season when compared to treatment with FLOVENT™ DISKUS™ 100 mcg.

DETAILED DESCRIPTION:
Study ADA113872 will assess the ability of ADVAIR™ DISKUS™ 100/50 mcg, in comparison to FLOVENT™ DISKUS™ 100 mcg, to reduce worsening asthma associated with viral respiratory infections during the fall season in a pediatric population. A number of descriptive measures will be used to assess the reduction in worsening asthma. These include the number of exacerbations, the duration and severity of asthma symptoms in the 7 days following the report of moderate upper respiratory tract symptoms or worsening asthma, the number of rescue-free days, and the rate of asthma control days.

Subjects will be identified starting in April 2010 to evaluate whether they meet the eligibility criteria. If a subject is identified as a potential candidate for the study they will be requested to return to the clinic between August 2, 2010 and August 20, 2010. Subjects who meet all inclusion and none of the exclusion criteria will be entered into the study. All subjects must be randomized on or before August 20th, 2010.

Subjects will be males and females who are between the ages of 4 and 11 years (as of randomization date) with a documented diagnosis of asthma requiring ICS monotherapy controller medication or low dose ICS as part of combination controller medication. In order for a subject on moderate dose ICS or low dose ICS + LABA combination therapy to be eligible for inclusion in this study their asthma must be under control for the 3 months prior to randomization and they must be a candidate for step-down therapy as outlined by current asthma management guidelines.

All subjects must have a history of one or more exacerbations during the previous respiratory viral season that required the use of outpatient oral/parenteral corticosteroid or an urgent care, Emergency Department visit hospitalization, or for asthma that required the use of oral/parenteral corticosteroid.

Subjects will receive their study medication at the Randomization visit and be instructed to keep an electronic daily record of AM PEF, asthma symptoms, night-time awakenings due to asthma, rescue use, and upper respiratory tract infection symptoms.

During the double-blind treatment period the electronic Diary (eDiary) will alert the subject or parent/legal guardian when the data imputed into the eDiary indicates the presence of upper respiratory symptoms of moderate or severe severity or if the subject has reached the criteria for worsening asthma. Upon receipt of either of these alerts, the subject or parent/legal guardian will be instructed to call the clinic. The clinic will instruct the subject (parent/legal guardian) to provide a mucus sample for assessment of viral respiratory infection. Mucus samples for viral respiratory assessment will not be collected from subjects more than once in a 7 day period. During the randomization visit subjects will receive training on the at home collection of a mucus sample.

Throughout the study each subject will be instructed to rate their daily upper respiratory symptoms. Upper respiratory tract symptoms include: runny nose, sneezing, nasal congestion, and sore throat. Subjects will be instructed to select a rating from the following list that best describes their aggregate upper respiratory symptoms during the previous 24 hours.

This study will evaluate the effects of the ADVAIR™ DISKUS™ 100/50 mcg and FLOVENT™ DISKUS™ 100 mcg on clinical parameters and indices of airway inflammation associated with viral respiratory tract infections in pediatric asthmatic subjects. Safety will be assessed by monitoring adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient
* Subjects must be between the ages of 4 and 11 at Randomization
* Subjects must attend day-care, pre-school, elementary school, or middle school. Day-care attendance is defined as receiving childcare outside the home for at least 10 hours per week. Children who are home-schooled are not eligible for this study. Children on year round and traditional school calendars are eligible for this study.
* Subjects can be randomized into this study at any time between August 2nd, 2010 and August 20th, 2010.
* Males or pre-menarchal females.
* A diagnosis of asthma, as defined by the National Institutes of Health [NIH, 2007]
* At Visit 1 subjects must demonstrate a best clinic AM PEF ≥70% of the predicted value [Polgar, 1971].
* Each subject must have a history of an exacerbation of asthma between September 1st, 2009 and May 15th, 2010 that required a burst of outpatient systemic corticosteroids (oral or parenteral on >1 days for worsening symptoms of asthma) or have had an urgent care, hospitalization, or ED visit for asthma during which they received oral/parenteral corticosteroids between September 1st, 2009 and May 15th, 2010.
* Subjects must have prior or current use of controller ICS medication as listed below:
* Subjects who have had prior use of a controller medication consisting of a low dose ICS at any time since September 1st, 2009 are eligible for inclusion in this study (refer to Table 1 for examples of allowed doses of commonly used ICS).
* Subjects currently taking a low dose ICS are eligible for inclusion in the study (refer to Table 1 for examples of allowed doses of commonly used ICS).
* Subjects' currently taking a moderate dose ICS are eligible for inclusion in the study if the subject's asthma has been controlled over the prior 3 months and the subject is a candidate for step down therapy, as defined by current asthma management guidelines [NIH, 2007].
* Subjects' currently taking low dose ICS in combination with a LABA are eligible for inclusion in the study if the subject's asthma has been controlled over the prior 3 months and the subject is a candidate for step down therapy, as defined by current asthma management guidelines [NIH, 2007].
* All subjects must be able to replace their short-acting beta2-agonists with study-issued albuterol inhalation aerosol at Visit 1 for use as needed for the duration of the study. If a subject demonstrates the inability to coordinate the use of an MDI alone, subjects are permitted to use an Aerochamber Plus spacer. The use or non-use of a spacer for albuterol inhalation aerosol should be consistent for each subject throughout the study. Subjects must be able to withhold inhaled albuterol for at least 6 hours prior to study Visits
* Chickenpox: Reported history of clinical varicella or varicella vaccine. If a subject needs varicella vaccine this will be arranged with a physician and must be received prior to randomization.
* Electronic Peak Flow Meter (ePEF)/Electronic Daily Diary (eDiary): A subject must be able to use the study-provided electronic peak flow meter and the subject/caregiver must be able to enter data using the electronic Diary record.
* Responsibilities of Consenting Parent/Legal Guardian: The subject's parent or legal guardian must commit to assist the subject at a consistent level with administration of investigational product and electronic Diary device and electronic PEF meter throughout the study.
* A subject must demonstrate adequate and appropriate technique for using the DISKUS™ device reliably.
* Fluency in English or USA Spanish: Subject and/or subject's parent/guardian must be able to read, comprehend, and record information in English or USA Spanish.

Exclusion Criteria:

* History of Life Threatening Asthma
* Unstable Asthma
* Concomitant use of corticosteroid medication
* Other Concurrent Diseases/Abnormalities: The known presence of sinus, middle ear, oropharyngeal, upper or lower respiratory tract infections within 4 weeks immediately preceding randomization that required the use of an antibiotic or was accompanied by symptoms of worsening asthma.
* Concomitant Medications: Administration of any other prescription or over the counter medication which would significantly affect the course of asthma, such as omalizumab (Xolair), or interact with sympathomimetic amines, such as: anticonvulsants (barbiturates, hydantoins, carbamazepine), polycyclic antidepressants, beta-adrenergic blocking agents (both cardio-selective and non-selective), phenothiazines,
* Cytochrome P450 3A4 (CYP 3A4) Inhibitors: A subject is not eligible if he/she is receiving a strong CYP 3A4 inhibitor within 4 weeks of Visit 1 (e.g., ritonavir, ketoconazole, itraconazole).
* Immunosuppressive medications: A subject must not be using or require use of immunosuppressive medications (e.g. methotrexate, gold, cyclosporine, azathioprine) during the study.

Note: Immunotherapy for the treatment of allergies is allowed during the study provided it was initiated 4 weeks prior to Visit 1 and the subject remains in the maintenance phase for the duration of the study.

* Concurrent Respiratory Disease: A subject must not have current evidence of pneumonia, pneumothorax, atelectasis, pulmonary fibrotic disease, bronchopulmonary dysplasia, chronic bronchitis, emphysema, cystic fibrosis, dyspnea by any cause other than asthma, or other respiratory abnormalities other than asthma.
* Other Concurrent Diseases/Abnormalities: Historical or current evidence of clinically significant uncontrolled disease that in the opinion of the investigator would put the safety of the subject at risk through study participation or would confound the interpretation of the results if the condition/disease exacerbated during the study.

The list of additional excluded conditions/diseases includes, but is not limited to the following:

Uncontrolled hypertension; Uncontrolled hematologic, hepatic, neurologic, or renal disease Uncontrolled gastroesophageal reflux disease, Immunologic compromise, Cardiac arrhythmias, Tuberculosis (current or untreated), Congestive heart failure, Cushing's disease Coronary artery disease, Addison's disease, Current malignancy, Eosinophilic esophagitis Uncontrolled diabetes mellitus, Uncontrolled thyroid disorder

* Severe Hypersensitivity to Milk Proteins: Any immediate hypersensitivity reaction, such as urticaria, angioedema, rash, and bronchospasm to milk proteins
* Drug Allergy: Any adverse reaction including immediate or delayed hypersensitivity to any beta2-agonist, sympathomimetic drug, or any intranasal, inhaled or systemic corticosteroid therapy. Known or suspected sensitivity to the constituents of the Dry Powder Inhaler (i.e., lactose).
* Tobacco Use: A history of or present use of any tobacco products.
* Investigational Medications: A subject must not have participated in a study (including a non-interventional study) or used any investigational drug (including devices) within 30 days prior to Visit 1 or within ten half-lives (t1/2) of the prior investigational study (whichever is longer of the two).
* Child in Care: A Child in Care (CiC) is a child who has been placed under the control or protection of an agency, organisation, institution or entity by the courts, the government or a government body, acting in accordance with powers conferred on them by law or regulation. The definition of a CiC can include a child cared for by foster parents or living in a care home or institution, provided that the arrangement falls within the definition above. The determination of whether a child meets the definition of CiC should be made with the study centre staff in consultation with the responsible IRB/Ethics Committee.
* Affiliation with Investigator's Site: A subject is an immediate family member of the participating investigator, sub investigator, study coordinator, or employee of the participating investigator.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 339 (Actual)
Dates: Start 2010-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (36):
- United States (36):
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Granada Hills, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Gainesville, Georgia
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Owensboro, Kentucky
  - GSK Investigational Site, Ypsilanti, Michigan
  - GSK Investigational Site, Brick, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Collegeville, Pennsylvania
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Summerville, South Carolina
  - GSK Investigational Site, Boerne, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, Murray, Utah
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Prazma CM, Gern JE, Weinstein SF, Prillaman BA, Stempel DA. The association between seasonal asthma exacerbations and viral respiratory infections in a pediatric population receiving inhaled corticosteroid therapy with or without long-acting beta-adrenoceptor agonist: a randomized study. Respir Med. 2015 Oct;109(10):1280-6. doi: 10.1016/j.rmed.2015.06.010. Epub 2015 Jun 24. PMID 26289742
- See also: National Health Lung and Blood Institute Asthma Guidelines — http://www.nhlbi.nih.gov/guidelines/asthma/
- Available data/document: Informed Consent Form: 113872 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113872 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113872 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113872 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113872 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113872 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113872 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- FSC DISKUS 100/50 mcg BID: Fluticasone Propionate/Salmeterol DISKUS Combination Product (FSC) at a dose of 100/50 micrograms (mcg) administered as one inhalation twice daily (BID) for 16 weeks
- FP DISKUS 100 mcg BID: Fluticasone Propionate (FP) DISKUS 100 mcg administered as one inhalation BID for 16 weeks
Period: Overall Study
Arm/Group | FSC DISKUS 100/50 mcg BID | FP DISKUS 100 mcg BID
Started | 171 | 168
Completed | 147 | 145
Not Completed | 24 | 23
Not completed — Withdrawal by Subject | 6 | 10
Not completed — Protocol Violation | 10 | 3
Not completed — Physician Decision | 2 | 4
Not completed — Lost to Follow-up | 3 | 3
Not completed — Adverse Event | 2 | 1
Not completed — Lack of Efficacy | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FSC DISKUS 100/50 mcg BID | FP DISKUS 100 mcg BID | Total
Number analyzed (Participants) | 171 | 168 | 339
Age, Continuous [Mean (Standard Deviation); unit: Years] | 7.5 (2.11) | 7.4 (2.08) | 7.4 (2.09)
Gender [Count of Participants; unit: Participants]
  Female | 63 | 56 | 119
  Male | 108 | 112 | 220
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 27 | 33 | 60
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 8 | 6 | 14
  American Indian or Alaska Native and White | 1 | 0 | 1
  White | 129 | 127 | 256
  African American/African Heritage and White | 1 | 1 | 2
  Asian & Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Asian and White | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander & White | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Asthma Exacerbations Reported During the Treatment Period
Description: An asthma exacerbation was defined as deterioration of asthma that required the use of outpatient oral/parenteral corticosteroids (tablets, suspensions, or injection) or an urgent care, hospitalization, or emergency room (ER) visit due to asthma that required oral/parenteral corticosteroids. Two exacerbations (out of a total of 51) were excluded: (1) one exacerbation occurred within 7 days of the resolution of an earlier one, and, per protocol, was combined with the previous exacerbation; and (2) one exacerbation occurred post treatment.
Time Frame: From Baseline (Week 1) until the end of treatment (up to Week 16)
Population: Intent-to-Treat (ITT) Population: all participants randomized to treatment. Only those participants who reported >=1 exacerbation were analyzed.
Measure: Number; unit: Number of asthma exacerbations
Arm/Group | FSC DISKUS 100/50 mcg BID | FP DISKUS 100 mcg BID
Number analyzed (Participants) | 21 | 20
Number of asthma exacerbations | 24 | 25
Statistical Analysis 1: Comparison: FSC DISKUS 100/50 mcg BID vs FP DISKUS 100 mcg BID; Test type: Superiority or Other; p = 0.928, Regression, Cox — Cox Proportional Hazards model adjusted for investigative center; Hazard Ratio (HR) = 0.971, 95% CI 2-sided [0.519 to 1.819] — The risk of having an asthma exacerbation during the treatment period was analyzed

2. Secondary Outcome: Mean Asthma Symptom Scores, as an Indicator of Severity, Associated With the Presence of Moderate or Severe Upper Respiratory Tract Symptoms (URTS) or a Confirmed Rhinovirus (RV) Infection at Baseline and During the Peak Viral Period
Description: Participants recorded their asthma symptom score over the previous 24 hours (during the day and the previous night) using the following 6-point scale: 0=No symptoms; 1=Symptoms for 1 short period; 2=Symptoms for >=2 short periods; 3=Symptoms for most of the day/previous night that did not affect normal daily activities; 4=Symptoms for most of the day/previous night that affected normal daily activities; 5=Symptoms so severe that participant could not perform normal daily activities. The Baseline mean asthma symptom score was calculated as the average score over 7 days prior to Week 1, Visit 2.
Time Frame: Baseline (Week 1) and Peak Viral Period ([period during which the greatest number of viral infections is expected] from 30 August 2010 through the end of the treatment period [up to Week 16])
Population: ITT Population. Only those participants with moderate or severe URTS or a confirmed RV infection were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- FSC DISKUS 100/50 mcg BID: FSC at a dose of 100/50 mcg administered as one inhalation BID for 16 weeks
- FP DISKUS 100 mcg BID: FP DISKUS 100 mcg administered as one inhalation BID for 16 weeks
Arm/Group | FSC DISKUS 100/50 mcg BID | FP DISKUS 100 mcg BID
Number analyzed (Participants) | 106 | 104
Scores on a scale
  Baseline, n=105, 104 | 0.2 (0.41) | 0.2 (0.39)
  Peak Viral Period, n=106, 104 | 0.5 (0.84) | 0.4 (0.70)

3. Secondary Outcome: Mean Duration of Worsening Asthma Symptoms Associated With the Presence of Moderate or Severe URTS or a Confirmed RV Infection
Description: A worsening asthma day is one on which any of the following occurred: rescue albuterol use above baseline, use of oral/parenteral corticosteroids for asthma, use of asthma medication other than study medication, asthma symptom scores >=3, nighttime awakenings, unscheduled health care visits, or missed school due to asthma. The duration of worsening asthma is the number of consecutive worsening asthma days after the date of a URTS score of 2 (moderate) or 3 (severe) or collection of a mucus sample containing RV (whichever occurred first). Each span of consecutive days is a participant interval.
Time Frame: Peak Viral Period (from 30 August 2010 through the end of treatment [up to Week 16])
Population: ITT Population. Only those participants with relevant data defining a worsening asthma day during the peak viral period and with moderate or severe URTS or a confirmed RV infection were analyzed.
Measure: Mean (Standard Error); unit: Days per participant interval
Arm/Group | FSC DISKUS 100/50 mcg BID | FP DISKUS 100 mcg BID
Number analyzed (Participants) | 121 | 145
Days per participant interval | 4.1 (0.18) | 4.0 (0.17)

4. Secondary Outcome: Number of Asthma Exacerbations Associated With the Presence of Moderate or Severe URTS or a Confirmed RV Infection During the Peak Viral Period
Description: Each participant (with assistance from the parent/legal guardian as needed) was instructed to keep an electronic diary (eDiary) with record of daily URTS symptoms that included: runny nose, sneezing, nasal congestion, and sore throat. Based on the best-described aggregate URTS during the previous 24 hours, participants rated symptoms as: 0 = Not present; 1 = Mild, clearly present; 2 = Moderately severe, uncomfortable; and 3 = Severe, interfering with sleep or activity. Mucus samples were collected and analyzed for RVwhen the eDiary alerted for moderate/severe URTS.
Time Frame: Peak Viral Period (from 30 August 2010 through the end of treatment [up to Week 16])
Population: ITT Population. Only those participants who reported >=1 exacerbation were analyzed. Only those participants with moderate or severe URTS or a confirmed RV infection were analyzed.
Measure: Number; unit: Number of asthma exacerbations
Arm/Group | FSC DISKUS 100/50 mcg BID | FP DISKUS 100 mcg BID
Number analyzed (Participants) | 5 | 7
Number of asthma exacerbations | 5 | 7

5. Secondary Outcome: Mean Percentage of Asthma-control Days
Description: An asthma-control day was defined as a day without any of the following: rescue albuterol use, use of oral/parenteral corticosteroids for asthma, use of asthma medication other than double-blind study treatment, asthma symptom score >0, nighttime awakenings due to asthma, unscheduled health care visits (defined as home visits, office visits, or urgent care visits), ER visits, hospitalizations for asthma, or school absenteeism due to asthma. The percentage of asthma-control days = the number (No.) of asthma-control days divided by the No. of days of treatment exposure, multiplied by 100.
Time Frame: Peak Viral Period (from 30 August 2010 through the end of treatment [up to Week 16])
Population: ITT Population. Only those participants who recorded data during the Peak Viral Period, had a treatment stop date with a defined Peak Viral Period, and had available data on all days on which data were recorded were analyzed.
Measure: Mean (Standard Error); unit: Percentage of days
Arm/Group | FSC DISKUS 100/50 mcg BID | FP DISKUS 100 mcg BID
Number analyzed (Participants) | 161 | 156
Percentage of days | 48.3 (1.51) | 49.7 (1.54)

6. Secondary Outcome: Mean Percentage of Episode-free (EF) Days
Description: An EF day was defined as a day without any of the following: rescue albuterol use, use of oral/parenteral corticosteroids for asthma, use of asthma medication other than study treatment, asthma symptom score >0, nighttime awakenings due to asthma, unscheduled health care visits (defined as home visits, office visits, or urgent care visits), ER visits, hospitalizations for asthma, school absenteeism due to asthma, or morning peak expiratory flow (measure of maximum airflow) <80% of baseline. Percentage of EF days=No. of EF days divided by No. of days of treatment exposure, multiplied by 100.
Time Frame: Peak Viral Period (from 30 August 2010 through the end of treatment [up to Week 16])
Population: as for outcome 5
Measure: Mean (Standard Error); unit: Percentage of days
Arm/Group | FSC DISKUS 100/50 mcg BID | FP DISKUS 100 mcg BID
Number analyzed (Participants) | 161 | 155
Percentage of days | 42.4 (1.55) | 44.5 (1.61)

7. Secondary Outcome: Mean Percentage of Symptom-free Days
Description: A symptom-free day was defined as a day during the Peak Viral Period on which the asthma symptom score was zero. The daily asthma symptom score (measured during the day and the previous night) was reported on a 6-point scale (ranging from 0=no symptoms to 5=severe symptoms). Percentage of symptom-free days was defined as the number of days during the Peak Viral Period on which the asthma symptom score=0, divided by the number of days in that same period on which non-missing values were recorded, multiplied by 100.
Time Frame: Peak Viral Period (from 30 August 2010 through the end of treatment [up to Week 16])
Population: ITT Population. Only those participants who recorded data during the Peak Viral Period and had a treatment stop date with a defined Peak Viral Period were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | FSC DISKUS 100/50 mcg BID | FP DISKUS 100 mcg BID
Number analyzed (Participants) | 161 | 157
Percentage of days | 90.1 (15.89) | 91.1 (13.18)

8. Secondary Outcome: Mean Percentage of Rescue-free Days
Description: A rescue-free day was defined as a day during the Peak Viral Period on which no puffs of rescue medication were recorded. Percentage of rescue-free days was defined as the number of days during the Peak Viral Period on which no puffs of rescue medication were recorded, divided by the number of days in that same period on which non-missing values were recorded, multiplied by 100.
Time Frame: Peak Viral Period (from 30 August 2010 through the end of treatment [up to Week 16])
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | FSC DISKUS 100/50 mcg BID | FP DISKUS 100 mcg BID
Number analyzed (Participants) | 161 | 157
Percentage of days | 92.1 (16.60) | 91.7 (14.68)

ADVERSE EVENTS:
Arm/Group | FSC DISKUS 100/50 mcg BID | FP DISKUS 100 mcg BID
Serious Adverse Events (participants affected / at risk) | 2/171 | 1/168
Other Adverse Events (participants affected / at risk) | 85/171 | 84/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FSC DISKUS 100/50 mcg BID (N=171) | FP DISKUS 100 mcg BID (N=168)
Gastroenteritis (Infections and infestations) | 1 | 0
Pneumonia respiratory syncytialviral (Infections and infestations) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FSC DISKUS 100/50 mcg BID (N=171) | FP DISKUS 100 mcg BID (N=168)
Upper respiratory tract infection (Infections and infestations) | 30 | 31
Nasopharyngitis (Infections and infestations) | 15 | 20
Sinusitis (Infections and infestations) | 11 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 26 | 21
Nasal congestion (Reproductive system and breast disorders) | 15 | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 | 12
Headache (Nervous system disorders) | 25 | 28
Pyrexia (General disorders) | 20 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.